CLINICAL TRIAL: NCT03811444
Title: Simulated Clinical Use Testing to Evaluate Sharps Injury Prevention Features of HTL-STREFA's Safety Lancets (Test A)
Brief Title: Simulated Clinical Use Testing On Safety Lancets (Test B)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HTL-Strefa S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Test B
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Needle Stick
Keywords: needlestick; needlestick injury; safety lancet; sharps injury prevention; capillary blood sampling
MeSH Terms: conditions — Needlestick Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- simulation of skin pricking type 420 (Experimental): The evaluator simulated the capillary blood sampling with the safety lancet type 420
  Interventions: Device: Haemolance Plus safety lancet
- simulation of skin pricking type 430 (Experimental): The evaluator simulated the capillary blood sampling with the safety lancet type 430
  Interventions: Device: Prolance safety lancet
- simulation of skin pricking type 520 (Experimental): The evaluator simulated the capillary blood sampling with the safety lancet type 520
  Interventions: Device: MediSafe Solo safety lancet

INTERVENTIONS:
Device: Haemolance Plus safety lancet — Haemolance Plus safety lancet type 420 is a sterile, single use medical device designed for the sampling of capillary blood from the fingertip of patients
  Arms: simulation of skin pricking type 420
Device: Prolance safety lancet — Prolance safety lancet type 430 is a sterile, single use medical device designed for the sampling of capillary blood from the fingertip of patients.
  Arms: simulation of skin pricking type 430
Device: MediSafe Solo safety lancet — MediSafe Solo safety lancet type 520 is a sterile, single use medical device designed for the sampling of capillary blood from the fingertip of patients.
  Arms: simulation of skin pricking type 520

SUMMARY:
A simulated clinical use testing on the HTL-Strefa's safety lancets

DETAILED DESCRIPTION:
This study aims to evaluate the safety of the use of the safety lancets: Haemolance Plus, Prolance and MediSafe Solo in the prevention of NSI and to evaluate the user's opinion with regards to the handling characteristics of the medical devices.

The simulated use clinical study will involve healthcare professionals (HCPs) who routinely use safety lancets to collect blood samples.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for HCP and lay person evaluators have been chosen based on FDA guidance:

* evaluators who routinely use safety lancets to collect capillary blood samples (prevention of the learning curve artifacts)
* evaluators will be United States (US) residents
* evaluators can read, write, and speak English
* evaluators are at least 18 years old
* evaluators are able to understand and provide signed consent for the study
* evaluators are willing to comply with the study protocol, including being willing to answer questions and complete questionnaires.
* evaluators have no concerns about the ability to perform the simulated skin pricking.

Exclusion Criteria:

Individuals will be excluded if:

* They do not routinely use safety lancets to collect capillary blood samples,
* They cannot read, write, and speak English,
* They or a family member have a business or consulting relationship with a pharmaceutical or medical device company, or
* They have participated in a product evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
The true failure rate of the tested devices | At time of testing, up to 90 minutes
Effectiveness of the safety lancet's sharps injury prevention features | At time of testing, up to 90 minutes
  Evaluator questionnaire using five-point response Likert scale (coded from 1 "strongly disagree" to 5 "strongly agree") to measure respondents' attitudes to a particular question or statement. Numbers assigned to Likert scale express a "greater than" relationship.

SECONDARY OUTCOMES:
Subjective assessments regarding evaluators' interactions with the tested safety lancets | At time of testing, up to 90 minutes
  Evaluator questionnaire using five-point response Likert scale (coded from 1 "strongly disagree" to 5 "strongly agree") to measure respondents' attitudes to a particular question or statement. Numbers assigned to Likert scale express a "greater than" relationship.
Safety of the devices based on the evaluators' assessments (five-point response scale) | At time of testing, up to 90 minutes
  Evaluator questionnaire using five-point response Likert scale (coded from 1 "strongly disagree" to 5 "strongly agree") to measure any and all observed needlestick injuries and device malfunctions. Numbers assigned to Likert scale express a "greater than" relationship.
Various aspects of the ease of use. | At time of testing, up to 90 minutes
  Evaluator questionnaire using five-point response Likert scale (coded from 1 "strongly disagree" to 5 "strongly agree") to measure respondents' attitudes to a particular question or statement. Numbers assigned to Likert scale express a "greater than" relationship.
Any handling, usability questions / issues associated with the device | At time of testing, up to 90 minutes
  Evaluator questionnaire using five-point response Likert scale (coded from 1 "strongly disagree" to 5 "strongly agree") to measure respondents' attitudes to a particular question or statement. Numbers assigned to Likert scale express a "greater than" relationship.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UL LLC, Chicago, Illinois
  - Schlesinger Associates, Boston, Massachusetts